CLINICAL TRIAL: NCT05842577
Title: Efficacy of Non-immersive Virtual Reality-based Telerehabilitation in Parkinson's Disease: a Multicentre Randomized Controlled Trial
Brief Title: RCT on Telerehabilitation Efficacy in Parkinson's Disease
Acronym: REPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Collaborators: Fondazione Don Carlo Gnocchi Onlus (Other); IRCCS National Neurological Institute "C. Mondino" Foundation (Other); Fondazione Salvatore Maugeri (Other); IRCCS San Camillo, Venezia, Italy (Other); IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP 01/18
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease
Keywords: Telerehabilitation; Parkinson; Balance; Continuity of Care
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This study is a multicentre, single-blind (evaluator), Randomized Controlled Trial (RCT)
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group (TG) (Experimental): The TG consisted of 30 sessions lasting approximately 45 minutes (3-5/week for 6-10 weeks) of motor, and cognitive rehabilitation exercises in non-immersive VR-based TR modality using the VRRS Tablet system (Khymeia Srl, Noventa Padovana, Italy).
  Interventions: Device: VRRS Tablet (Khymeia s.r.l., Noventa Padovana, Italy)
- Control Group (CG) (Active Comparator): The CG carried consisted of 30 sessions lasting approximately 45 minutes (3-5 days/week for, 6-10 weeks) of at-home conventional rehabilitation via structured self-administered exercises without the use of any technological devices.
  Interventions: Other: At-home conventional rehabilitation

INTERVENTIONS:
Device: VRRS Tablet (Khymeia s.r.l., Noventa Padovana, Italy) — The motor exercises were performed using inertial sensors for the acquisition and processing of the movement performed by the patient. The patient was trained to perform these exercises using visual and auditory feedback in a serious game environment. The exercises were aimed at the rehabilitation of balance and at the improvement of motor performance in lower limbs (e.g., maintaining balance on one leg, marching in place, standing on tiptoe, squatting, etc.). The therapists involved in the study customized the protocol of exercises in TR mode according to the characteristics and needs of the subject.
  Arms: Telerehabilitation Group (TG)
Other: At-home conventional rehabilitation — The CG rehabilitation was an active comparator treatment and consisted of a written home-based self-administered booklet with conventional motor activities tailored for each subject. The motor activities were chosen and adapted from a specialized manual. The motor exercises were aimed at the rehabilitation of balance and at the improvement of motor performance in lower limbs (e.g., maintaining balance on one leg, marching in place, standing on tiptoe, squatting, etc).
  Other Names: Structured self-administered exercises
  Arms: Control Group (CG)

SUMMARY:
The implementation of regular prolonged, and effective rehabilitation in people with Parkinson's disease is essential for ensuring a good quality of life. However, the continuity of rehabilitation care may find barriers related to economic, geographic, and social issues. In these scenarios, telerehabilitation could be a possible solution to guarantee the continuity of care.

This trial aims to investigate the efficacy of non-immersive virtual reality-based telerehabilitation on postural stability in people with Parkinson's disease, compared to at-home conventional rehabilitation.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a chronic degenerative pathology characterized by both motor and non-motor symptoms that may have a significant long-term impact on Activities of Daily Living (ADL).

Subjects with PD need continuous, intensive, and tailored rehabilitation in order to improve motor function as well as their Quality of Life (QoL), and to reduce the risk of balance impairment and falls. Thus, the implementation of regular prolonged, and effective rehabilitation in people with PD is essential for ensuring well-being.

In this scenario, the delivery of rehabilitation services at distance, namely TeleRehabilitation (TR), is a possible solution to guarantee the continuity of care and physical exercise at home via digital healthcare.

Although the TR intervention has been proposed as a sustainable and innovative approach in people with PD, there are still conflicting results in the literature about its efficacy.

This study aims to investigate the efficacy of non-immersive VR-based TR on postural stability in people with PD, compared to at-home conventional rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn & Yahr (H&Y) score between ≤3 (ON-state);
* the absence of moderate and severe dyskinesias assessed by the MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) with a score of items 4.1 and 4.2 < 3;
* the absence of moderate and severe freezing episodes assessed by the MDS-UPDRS with a score of items 2.13 and 3.11 < 3;
* the ability to perform the 6 Minutes Walking Test (6MWT) between 200 m and 600 m;
* age ≤ 80 years;
* the absence of cognitive impairment measured by the Montreal Cognitive Assessment (MoCA) total score≥17.54 ;
* stabilized drug treatment;
* sufficient cognitive and linguistic level to understand and comply with study procedures;
* sign informed consent.

Exclusion Criteria:

* other neurological pathologies, psychiatric complications, or personality disorders;
* blurred or low vision problems;
* hearing and speech impairment affecting participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the mini-Balance Evaluation Systems Test (mini-BESTest) | Session 1 (Baseline, T0), Session 30 (End of treatment, approximately 10 weeks, T1)]
  The mini-BESTest is a shortened version of the Balance Evaluation Systems Test. It aims to target and identify 6 different balance control systems so that specific rehabilitation approaches can be designed for different balance deficits. The test was shortened based on factor analysis to include dynamic balance only and to improve clinical utilization. It is 36 items scale that evaluates Balance with total score of 28.

SECONDARY OUTCOMES:
Change in the Timed Up and Go test (TUG) | Session 1 (Baseline, T0), Session 30 (End of treatment, approximately 10 weeks, T1)]
  The TUG test assesses mobility, balance, walking ability, and fall risk in older adults. It is a measure of function with correlates to balance and fall risk. The participant is asked to get up from the chair she/he is sitting in, walk the marked distance of 3 meters and return to her/his seat again. The elapsed time is recorded in seconds.
Change in the 6-minute WalkTest (6mWT) | Session 1 (Baseline, T0), Session 30 (End of treatment, approximately 10 weeks, T1)]
  The 6mWT assesses the functional exercise capacity. The patient is asked to walk as long as possible for 6 minutes at a self-selected speed. The distance is recorded in meters.
Change in the MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) - part III | Session 1 (Baseline, T0), Session 30 (End of treatment, approximately 10 weeks, T1)]
  MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. Part III assessed the motor signs of PD and was administered by the rater (Range 0-132). Part III contained 33 scores based on 18 items. For each question, a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. A higher score indicated more severe symptoms of PD.

CONTACTS AND LOCATIONS:
Overall Officials: Michela Goffredo, PhD, Principal Investigator — IRCCS San Raffaele Roma
Locations (6):
- Italy (6):
  - IRCCS Bonino-Pulejo, Messina
  - IRCCS Fondazione Don Carlo Gnocchi ONLUS, Milan
  - IRCCS Mondino Foundation, Pavia
  - IRCCS San Raffaele Roma, Rome
  - IRCCS San Camillo Hospital, Venice
  - ICS Maugeri SB IRCCS Veruno, Veruno

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vellata C, Belli S, Balsamo F, Giordano A, Colombo R, Maggioni G. Effectiveness of Telerehabilitation on Motor Impairments, Non-motor Symptoms and Compliance in Patients With Parkinson's Disease: A Systematic Review. Front Neurol. 2021 Aug 26;12:627999. doi: 10.3389/fneur.2021.627999. eCollection 2021. PMID 34512495
- [Background] Barbour PJ, Arroyo J, High S, Fichera LB, Staska-Pier MM, McMahon MK. Telehealth for patients with Parkinson's disease: delivering efficient and sustainable long-term care. Hosp Pract (1995). 2016;44(2):92-7. doi: 10.1080/21548331.2016.1166922. PMID 26982525
- [Background] Cikajlo I, Hukic A, Dolinsek I, Zajc D, Vesel M, Krizmanic T, Blazica B, Biasizzo A, Novak F, Peterlin Potisk K. Can telerehabilitation games lead to functional improvement of upper extremities in individuals with Parkinson's disease? Int J Rehabil Res. 2018 Sep;41(3):230-238. doi: 10.1097/MRR.0000000000000291. PMID 29757774